CLINICAL TRIAL: NCT00723047
Title: Fibrin Glue for Perianal Fistulas in Crohn's Disease: a Randomized Controlled Trial
Acronym: Fibrin glue
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe d'Etude Therapeutique des Affections Inflammatoires Digestives (Other)
Collaborators: Nycomed (Industry); Société Nationale Française de Gastroentérologie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GETAID 2003-1
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Last update posted 2011-09-05 (Estimated); Status verified 2011-09

CONDITIONS: Crohn's Disease
Keywords: Patients; CD complicated; least; One perianal fistula; Draining; 2 months duration
MeSH Terms: conditions — Crohn Disease | interventions — Fibrin Tissue Adhesive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: Fibrin glue injection in fistula

INTERVENTIONS:
Procedure: Fibrin glue injection in fistula

SUMMARY:
This multicenter, randomized, controlled trial was conducted by the Groupe d'Etude Thérapeutique des Affections Inflammatoires du tube Digestif (GETAID) to evaluate the efficacy and safety of the injection of fibrin glue in perianal fistulas tracts of patients with CD. The institutional Independent Ethics Committee of Marseille, France and of Liège, Belgium approved the protocol for each participating centers. Recruitment took place at 12 sites (11 in France and 1 in Belgium)

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* CD confirmed by endoscopy and histology.
* CDAI should be 250 or less
* at least one perianal fistula (between anus or low rectum and perineum, vulva or vagina) draining for more than 2 months duration

Exclusion Criteria:

* treatment with an anti-TNF agent or with ciclosporin or tacrolimus within the last 3 months
* presence of a perianal abscess (>1cm) assessed by magnetic resonance imaging (MRI) or endo-anal ultrasonography performed within the last month,
* presence of anal or rectal stenosis,
* surgery during the previous month (except seton removal),
* previous fibrin glue injection,
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2003-11; Primary Completion 2006-06 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Clinical Remission | 8 weeks after inclusion
  Clinical remission was defined as
  * the absence of any draining by fistula openings occurring spontaneously or after gentle finger compression ,
  * the absence of perianal pain
  * and the absence of perianal abscess.

SECONDARY OUTCOMES:
Early Clinical Remission | 4 weeks after Inclusion
Occurrence of perianal abcess | During whole study

CONTACTS AND LOCATIONS:
Locations (14):
- Sart Tilman University Hospital, Liège, Belgium
- France (13):
  - Beaujon Hospital, Clichy
  - Louis Mourrier Hospital, Colombes
  - CHRU Lille, Lille
  - Marseille North Hospital, Marseille
  - Nice University Hospital, Nice
  - Hopital St Louis, Paris
  - Lariboisiere Hospital, Paris
  - Georges Pompidou European Hospital, Paris
  - Bichat Hospital, Paris
  - Lyon Sud University Hospital, Pierre-Bénite
  - Pontchaillou University Hospital, Rennes
  - Rouen University Hospital, Rouen
  - Trousseau University Hospital, Tours

REFERENCES:
- [Background] Hellers G, Bergstrand O, Ewerth S, Holmstrom B. Occurrence and outcome after primary treatment of anal fistulae in Crohn's disease. Gut. 1980 Jun;21(6):525-7. doi: 10.1136/gut.21.6.525. PMID 7429313
- [Background] Schwartz DA, Loftus EV Jr, Tremaine WJ, Panaccione R, Harmsen WS, Zinsmeister AR, Sandborn WJ. The natural history of fistulizing Crohn's disease in Olmsted County, Minnesota. Gastroenterology. 2002 Apr;122(4):875-80. doi: 10.1053/gast.2002.32362. PMID 11910338
- [Background] Schwartz DA, Pemberton JH, Sandborn WJ. Diagnosis and treatment of perianal fistulas in Crohn disease. Ann Intern Med. 2001 Nov 20;135(10):906-18. doi: 10.7326/0003-4819-135-10-200111200-00011. PMID 11712881
- [Background] Bernstein LH, Frank MS, Brandt LJ, Boley SJ. Healing of perineal Crohn's disease with metronidazole. Gastroenterology. 1980 Aug;79(2):357-65. PMID 7399243
- [Background] Present DH, Korelitz BI, Wisch N, Glass JL, Sachar DB, Pasternack BS. Treatment of Crohn's disease with 6-mercaptopurine. A long-term, randomized, double-blind study. N Engl J Med. 1980 May 1;302(18):981-7. doi: 10.1056/NEJM198005013021801. PMID 6102739
- [Background] Pearson DC, May GR, Fick GH, Sutherland LR. Azathioprine and 6-mercaptopurine in Crohn disease. A meta-analysis. Ann Intern Med. 1995 Jul 15;123(2):132-42. doi: 10.7326/0003-4819-123-2-199507150-00009. PMID 7778826
- [Derived] Grimaud JC, Munoz-Bongrand N, Siproudhis L, Abramowitz L, Senejoux A, Vitton V, Gambiez L, Flourie B, Hebuterne X, Louis E, Coffin B, De Parades V, Savoye G, Soule JC, Bouhnik Y, Colombel JF, Contou JF, Francois Y, Mary JY, Lemann M; Groupe d'Etude Therapeutique des Affections Inflammatoires du Tube Digestif. Fibrin glue is effective healing perianal fistulas in patients with Crohn's disease. Gastroenterology. 2010 Jun;138(7):2275-81, 2281.e1. doi: 10.1053/j.gastro.2010.02.013. Epub 2010 Feb 20. PMID 20178792
- See also: Related Info — http://www.getaid.org